CLINICAL TRIAL: NCT02257450
Title: Primary Aldosteronism in Malaysia: A Nationwide Multicentre Study
Acronym: MyEndo-PA
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: International Islamic University Malaysia (Other)
Collaborators: Malaysian Endocrine and Metabolic Society (Other); National University of Malaysia (Other); University of Malaya (Other); IMU University, Malaysia (Other)
Responsible Party: Principal Investigator, Dr Mohamnmad Arif Shahar, Assist Prof, International Islamic University Malaysia
Other Study IDs: MyEndo - PA
Record Dates: First submitted 2014-10-02; First posted 2014-10-06 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: Primary Aldosteronism
Keywords: Primary Aldosteronism; Hyperaldosteronism
MeSH Terms: conditions — Hyperaldosteronism

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum, plasma
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This research focuses on the prevalence of Primary Aldosteronism in the Malaysian adult population.

DETAILED DESCRIPTION:
Hypertension (HPT) is a very common disease, expensive to treat with serious morbidity and mortality. In Malaysia, from the NHMS III conducted in 2006, HPT affects more than 36% of adults. Essential HPT (HPT with no identifiable cause) accounts for approximately 85% of cases, whereas 15% have identifiable conditions (secondary cause). The detection of a secondary cause of HPT is important as the condition is reversible when detected early. Primary aldosteronism (PA) has been identified as the commonest cause of secondary HPT. At present, PA has been regarded as the commonest and potentially curable, with a prevalence of 5-13% [1-7]. If this condition is detected early, the chances of cure from hypertension have been reported up to 80% of cases.

This will translate to a major impact to the Malaysian health-care budget. The costs spent on life-long BP medications and complications related to HPT can be reduced enormously. PA is a type of hormonal disorder that leads to high blood pressure (BP). In PA, the adrenal glands produce too much aldosterone causing sodium retention and potassium excretion. The excess sodium then increased the blood volume and BP.

Diagnosis and treatment of this condition are of paramount importance because people with this form of high BP have a higher risk of heart attack, stroke, kidney impairment, metabolic abnormality and reduce quality of life compared to patients with high BP not due to this condition. More importantly, the high BP associated with PA may be curable. This research will be conducted as a multicenter nation-wide study in Malaysia. The research aimed to study the prevalence of this disease in the investigators Malaysian population, determine the underlying mechanisms why this disease is associated with higher complication rate through cardiovascular and inflammatory markers, and identify the genes causing this disease, hence provide a more rapid diagnostic test and possibility of curing the disease with genetic therapy

ELIGIBILITY:
Inclusion Criteria:

* 18 years old and above
* Malaysian citizen
* Consent given

Exclusion Criteria:

* Those who refused consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Malaysian adult population
Sampling Method: Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2014-10; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Aldosterone-Renin Ratio | Day 0
  Aldosterone-renin ratio of respondent at the time of sampling

SECONDARY OUTCOMES:
Level of Inflammatory Markers | Day 0
  Level of inflammatory markers (IL-6, hs-CRP) among respondents at the time of sampling
Level of cardiovascular markers | Day 0
  Level of cardiovascular markers (BNP, PAI-1) among respondents at the time of sampling

CONTACTS AND LOCATIONS:
Overall Officials: Nor Azmi Kamaruddin, FACE, Principal Investigator — Malaysian Endocrine and Metabolic Society